CLINICAL TRIAL: NCT00774475
Title: Optimization of Antiplatelet Therapy With Clopidogrel on the Basis of the Extent of Platelet Inhibition in Patients With Acute Coronary Syndromes on Dual Antiplatelet Therapy Undergoing PCI With Stent Implantation
Brief Title: Dual Antiplatelet Therapy Tailored on the Extent of Platelet Inhibition
Acronym: DANTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Florence (Other)
Collaborators: Tuscany Region (Unknown)
Responsible Party: Gian Franco Gensini, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Unstable Angina; NSTEMI
Keywords: Clopidogrel therapy; platelet function inhibition
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: standard therapy (Placebo Comparator): clopidogrel 75 mg/day
  Interventions: Drug: comparison of different dosage of clopidogrel
- 2: doubled therapy (Active Comparator): clopidogrel 150 mg/day
  Interventions: Drug: doubled therapy

INTERVENTIONS:
Drug: comparison of different dosage of clopidogrel — clopidogrel 75 mg/day versus clopidogrel 150 mg/day
  Arms: 1: standard therapy
Drug: doubled therapy — clopidogrel 150 mg/day
  Arms: 2: doubled therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy (reduction of major ischemic events at 6 and 12 months of follow-up) of a tailored clopidogrel therapy in patients with UA/NSTEMI undergoing PCI with stent implantation and wiht a documented residual platelet reactivity assessed by a point of care system (VerifyNow P2Y12).

DETAILED DESCRIPTION:
Several studies documented the presence of a high variability in the individual response to antiplatelet therapies in terms of extent of platelet function inhibition. This laboratory finding is the so-called aspirin or clopidogrel resistance which we prefer to define residual platelet reactivity (RPR) on antiplatelet therapy.

A growing body of evidence is demonstrating the clinical relevance of this laboratory parameter, i.e. patients with RPR are at higher risk of a subsequent adverse cardiovascular event.

In particular, it has been demonstrated that RPR measured by light transmittance aggregometry induced by ADP or by the point of care assay VerifyNow P2Y12 identifies patients which, after coronary revascularization with stent implantation, at higher risk of a potentially catastrophic event such as stent thrombosis.

No randomized trials are available in the literature on the efficacy and safety of an antiplatelet therapy tailored on the extent of platelet function inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Unstable or NSTEMI

Exclusion Criteria:

Previous bleeding events which have required blood transfusion

* PT- INR >1.5
* Platelet count ≤ 100000/ mm3
* Hb < 10 g/dl
* Previous TIA/stroke (ischemic or hemorrhagic or unknown)
* Body weight < 60 Kg
* Creatinine levels ≥ 4 mg/dl
* Cerebral neoplasia
* Recent major trauma/surgery/head injury (within 3 previous weeks)
* Gastrointestinal hemorrhage in the last month
* Aortic dissection
* Known haemorrhagic diathesis
* Oral anticoagulant therapy
* Pregnancy or 1 week after delivery
* Uncontrolled hypertension (systolic >180 mmHg or diastolic >110 mmHg)
* Severe liver disease
* Infective endocarditis
* Major psychiatric disorders
* Alcool or drug abuse
* Active peptic ulcer Noncompressible arterial puncture within 14 days Prolonged cardiopulmonary resuscitation

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE (cardiovascular death, nonfatal myocardial infarction, target lesion vessel revascularization by PCI or coronary bypass) | 6 and 12 months

SECONDARY OUTCOMES:
Stent thrombosis with angiographic confirmation; platelet function assessed by VerifyNow P2Y12 1 week after the randomization | 1 week; 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gian Franco Gensini, MD, Principal Investigator — University of Florence; Gianni Maria Santoro, MD, Study Chair — ASL 10 Florence, Italy; Niccolò Marchionni, MD, Study Chair — University of Florence; David Antoniucci, MD, Study Chair — Azienda Ospedaliero-Universitaria Careggi; Alfredo Zuppiroli, MD, Study Chair — ASL 10 Florence Italy; Maria Cristina Landini, MD, Study Chair — ASL 10 Florence Italy; Rosanna Abbate, MD, Study Director — University of Florence
Locations (1):
- University of Florence, Florence, Italy

REFERENCES:
- [Background] Gori AM, Marcucci R, Migliorini A, Valenti R, Moschi G, Paniccia R, Buonamici P, Gensini GF, Vergara R, Abbate R, Antoniucci D. Incidence and clinical impact of dual nonresponsiveness to aspirin and clopidogrel in patients with drug-eluting stents. J Am Coll Cardiol. 2008 Aug 26;52(9):734-9. doi: 10.1016/j.jacc.2008.05.032. PMID 18718420
- [Background] Buonamici P, Marcucci R, Migliorini A, Gensini GF, Santini A, Paniccia R, Moschi G, Gori AM, Abbate R, Antoniucci D. Impact of platelet reactivity after clopidogrel administration on drug-eluting stent thrombosis. J Am Coll Cardiol. 2007 Jun 19;49(24):2312-7. doi: 10.1016/j.jacc.2007.01.094. Epub 2007 Jun 4. PMID 17572245
- [Background] Price MJ, Endemann S, Gollapudi RR, Valencia R, Stinis CT, Levisay JP, Ernst A, Sawhney NS, Schatz RA, Teirstein PS. Prognostic significance of post-clopidogrel platelet reactivity assessed by a point-of-care assay on thrombotic events after drug-eluting stent implantation. Eur Heart J. 2008 Apr;29(8):992-1000. doi: 10.1093/eurheartj/ehn046. Epub 2008 Feb 10. PMID 18263931
- [Background] Santoro GM, Carrabba N, Barchielli A, Balzi D, Marchionni N, Filice M, Valente S, Granelli M, Berni I, Buiatti E; AMI-Florence Working Group. Use and efficacy of abciximab in an unselected population with acute myocardial infarction treated with primary angioplasty: data from AMI-Florence registry. Atherosclerosis. 2007 Nov;195(1):116-21. doi: 10.1016/j.atherosclerosis.2006.08.053. Epub 2006 Sep 25. PMID 16997308
- [Background] Balzi D, Barchielli A, Buiatti E, Franceschini C, Lavecchia R, Monami M, Santoro GM, Carrabba N, Margheri M, Olivotto I, Gensini GF, Marchionni N; AMI-Florence Working Group. Effect of comorbidity on coronary reperfusion strategy and long-term mortality after acute myocardial infarction. Am Heart J. 2006 May;151(5):1094-1100. doi: 10.1016/j.ahj.2005.06.037. PMID 16644342